CLINICAL TRIAL: NCT05641753
Title: CHORD1 - CHOlesterol Lowering and Residual Risk in Diabetes, Type 1
Brief Title: Cholesterol Lowering and Residual Risk in Diabetes, Type 1
Acronym: CHORD1
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-01095
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — evolocumab; Atorvastatin; Ezetimibe; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- 4-Week LDL-Cholesterol (LDL-C)-Reduction Treatment (Experimental): Treatment consists of: Evolocumab (140 mg; 2 injections, one administered at baseline visit and another self-administered 2 weeks later), and; Atorvastatin (up to 80mg dose; 1 tab per day for 30 days, starting at baseline visit post-assessment). Participants with statin intolerance will be provided with a 1-month supply of ezetimibe 10 mg to replace Evolocumab and Atorvastatin.
  * Additional procedures: Blood draws.
  * Optional procedures: Glycocalyx testing, PET/CT, or Endothelial Cell Collection.
  Interventions: Drug: Evolocumab Cartridge; Drug: Atorvastatin Calcium Tablets; Drug: Ezetimibe Tablets; Drug: 18F-FDG; Device: Angiocatheter 20IV; Device: J-Wire; Device: GlycoCheck Glycocalyx Measurement Software

INTERVENTIONS:
Drug: Evolocumab Cartridge — Injectable PCSK9 inhibitor.
  Other Names: REPATHA
Drug: Atorvastatin Calcium Tablets — HMG-CoA reductase inhibitor for oral use.
  Other Names: LIPITOR
Drug: Ezetimibe Tablets — Will only be distributed to patients with statin intolerance; replacement for both Atorvastatin and Evolocumab. Inhibitor of intestinal cholesterol for oral use.
  Other Names: ZETIA
Drug: 18F-FDG — Optional procedure. Positron emission tomography (PET) and computed tomography (CT) imaging to assess vascular inflammation and related anatomy requires injection of the PET tracer 18F-FDG. 18F-FDG is an FDA-approved analogue of sugar, routinely used to evaluate elevated metabolism in tissues, including increased metabolism due to inflammatory cells. A standard dose of 7.0 mSv will be administered.
Device: Angiocatheter 20IV — Optional procedure (endothelial cell harvesting). An angiocatheter ≤ 21 gauge will be inserted into a peripheral vein on the upper extremity using aseptic technique. A 0.018in. diameter J-shaped wire (Arrow, Reading, PA) will be then advanced into the angiocatheter, to a distance of 4cm beyond the end of the angiocatheter.
  Other Names: BD Insyte Autoguard
Device: J-Wire — Optional procedure (endothelial cell harvesting). Either a 0.021in. diameter J-shaped wire (Daig, Minnetonka, MN) or a 0.018in. diameter J-shaped wire (Arrow, Reading, PA) will be used.
Device: GlycoCheck Glycocalyx Measurement Software — Optional procedure (assessment of vascular function). Video microscope developed by GlycoCheck.

SUMMARY:
This is a prospective, interventional, cohort study, meaning that researchers will follow and observe a group of enrolled study participants over a period of time (one to two months) to gather information and record any developments of the outcomes in question.

This study will recruit 125 participants with Type 1 Diabetes (T1D) to:

1. Analyze the effect of reducing the cholesterol levels in the blood on platelet function. (Platelets are small cells in the blood which help form blood clots to slow or stop bleeding and to help wounds heal
2. Analyze the effect of reducing the cholesterol levels in the blood on While Blood Cell (WBC) gene expression, (White Blood Cells are part of the body's immune system which help the body fight infection and other diseases) and
3. Analyze the effect of reducing the cholesterol levels in the blood on vascular or blood vessel function.

DETAILED DESCRIPTION:
Participants will receive weekly injections of PCSK9i (evolocumab) plus daily, oral pills of atorvastatin or ezetimibe for 1 month.

Participants will undergo blood draw, and optional vascular studies that include:

* Glycocalyx testing (A non-invasive test where a video microscope camera is placed under the tongue to capture images of the movement of red blood cells as they travel through the micro-blood vessels)
* PET/CT for vascular imaging - to assess any inflammation of blood vessels and to evaluate increased metabolism in related tissues, and
* Endothelial cell collection before cholesterol reduction and 1-month after cholesterol reduction to measure any genetic changes in in the endothelial cells before and after collection

Glycemic Variability (GV), the amount one's blood sugar changes throughout the day, will be analyzed from continuous glucose monitoring (CGM) data.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with previous diagnosis of T1D (as defined by American Diabetes Association or judgment of physician for at least 1 year)

   1. American Diabetes Association Criteria for diagnosis of diabetes (Must meet at least 1 of the following criteria):

      * i. FPG ≥126 mg/dL (7.0 mmol/L). Fasting is defined as no caloric intake for at least 8 hours, OR;
      * ii. 2-h PG ≥200 mg/dL (11.1 mmol/L) during OGTT. The test should be performed using a glucose load containing the equivalent of 75 g anhydrous glucose dissolved in water, OR;
      * iii. A1C ≥6.5% (48 mmol/mol), OR;
      * iv. In a patient with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose ≥200 mg/dL (11.1 mmol/L), AND;
   2. History of T1D (due to autoimmune β-cell destruction, usually leading to absolute insulin deficiency, including latent autoimmune diabetes of adulthood). Autoimmune markers include islet cell autoantibodies and autoantibodies to GAD (glutamic acid decarboxylase, GAD65), insulin, the tyrosine phosphatases islet antigen 2 (IA-2) and IA-2β, and zinc transporter 8, OR;
   3. Diagnosis of T1D and confirmed by review of records by 2 separate clinical members of the study team
2. Age ≥ 18 & < 90
3. LDL-C >100mg/dl
4. Able and willing to provide written informed consent for the study

Exclusion Criteria:

1. Established cardiovascular disease on antithrombotic therapy
2. Triglycerides >400mg/dl
3. Use of a PCSK9 inhibitor
4. Recent infection in the past 30 days
5. Any hospitalization in the past 30 days
6. Use of immunosuppressive therapy
7. Use of any antithrombotic therapy
8. Use of aspirin
9. Use of NSAID within the past 72 hours
10. Pregnancy
11. Anemia (hemoglobin < 9 g/dl) or thrombocytopenia (platelet count <75), or thrombocytosis (platelet count >600)
12. A history of hemorrhagic diathesis
13. Chronic kidney disease (CrCl < 30ml/min)
14. T2D, monogenic diabetes syndromes, or diabetes in the context of disease of the exocrine pancreas (such as pancreatitis, trauma or pancreatectomy, neoplasia, cystic fibrosis, hemochromatosis)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Monocyte Platelet Aggregation (MPA) from Baseline | Baseline, Week 4
  Measurement of platelet activity. Assessed via patient blood sample.
Change in Light Transmission Aggregation (LTA) from Baseline | Baseline, Week 4
  Measurement of platelet activity. Assessed via patient blood sample.

SECONDARY OUTCOMES:
Percent Change in Natural Killer (NK) Cell Population from Baseline | Baseline, Week 4
  Assessed via patient blood sample.
Percent Change in Dendritic Cell Population from Baseline | Baseline, Week 4
  Assessed via patient blood sample.
Percent Change in CD8 Cell Population from Baseline | Baseline, Week 4
  Assessed via patient blood sample.

CONTACTS AND LOCATIONS:
Overall Officials: Ira Goldberg, MD, Principal Investigator — NYU Langone Health
Locations (4):
- United States (4):
  - New York VA Hospital, New York, New York
  - NYC Health + Hospitals/Bellevue, New York, New York
  - NYU Langone Health, New York, New York
  - Mount Sinai School of Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, will be shared upon reasonable request beginning immediately following publication provided the researchers who provide a methodologically sound proposal for use of the data execute a data use agreement with NYU Langone Health. Requests should be directed to Ira.Goldberg@nyulangone.org. The protocol, statistical analysis plan, informed consent form, clinical study report, and analytic code will be made available on Clinicaltrials.gov.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal will have access to the data upon reasonable request. Requests should be directed to Ira.Goldberg@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.